CLINICAL TRIAL: NCT05887843
Title: An Open-label, Single-Dose, Three-way Crossover Study to Compare the Pharmacokinetics of Fixed-Dose Combination of Mometasone + Azelastine Nasal Spray to Mometasone and Azelastine Nasal Sprays in Adolescents (12 to 17 Years of Age) and Young Adults (18 to 24 Years of Age) With Seasonal Allergic Rhinitis
Brief Title: Study to Compare the Pharmacokinetics of Fixed-Dose Combination of Mometasone + Azelastine Nasal Spray to Mometasone and Azelastine Nasal Sprays in Adolescents and Young Adults With Seasonal Allergic Rhinitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision (no safety concerns).
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SAN-0791; 2023-000362-34 (EudraCT Number)
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Mometasone Furoate; azelastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mometasone + Azelastine, then Mometasone Furoate, then Azelastine Hydrochloride (Experimental)
  Interventions: Drug: Mometasone + Azelastine; Drug: Mometasone Furoate; Drug: Azelastine Hydrochloride
- Mometasone Furoate, then Azelastine Hydrochloride, then Mometasone + Azelastine (Experimental)
  Interventions: Drug: Mometasone + Azelastine; Drug: Mometasone Furoate; Drug: Azelastine Hydrochloride
- Azelastine Hydrochloride, then Mometasone + Azelastine, then Mometasone Furoate (Experimental)
  Interventions: Drug: Mometasone + Azelastine; Drug: Mometasone Furoate; Drug: Azelastine Hydrochloride

INTERVENTIONS:
Drug: Mometasone + Azelastine — Mometasone + Azelastine, 50 μg/140 μg (per actuation) liquid, nasal spray, two actuations administered in each nostril
Drug: Mometasone Furoate — Mometasone Furoate 50 μg (per actuation) nasal spray, two actuations administered in each nostril
Drug: Azelastine Hydrochloride — Azelastine Hydrochloride 140 μg (per actuation) nasal spray, two actuations administered in each nostril

SUMMARY:
This study will compare the PK parameters of the combination test formulation to monotherapy reference products (mometasone furoate and azelastine hydrochloride) in adolescents and young adult patients with seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking, adolescent or young adult male and female subjects with seasonal allergic rhinitis.
2. Willing to use acceptable, effective methods of contraception.
3. Be informed of the nature of the study and give written consent (adults) / assent and consent by legal guardian(s)/parent(s) (adolescents) prior to any study procedure.

Exclusion Criteria:

1. Known history or presence of clinically significant disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. Known history or presence of hypersensitivity or idiosyncratic reaction to mometasone, azelastine, or any other drug substances with similar activity.
3. Unable to tolerate direct venipuncture.
4. Positive test result for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
5. Positive test result for urine drugs of abuse or urine cotinine.
6. Presence of nostril or septum piercing.
7. Use of tobacco or nicotine-containing products within 6 months prior to drug administration.
8. Females who are pregnant, breast-feeding, or have used hormonal contraceptives within 21 days (oral and transdermal) or 6 months (implanted, injected, intravaginal, or intrauterine) prior to drug administration.
9. Donation or loss of whole blood (including clinical trials) within 30 days prior to drug administration (or 56 days for ≥500 mL).
10. Participation in a clinical trial that involved administration of an investigational medicinal product within 30 days prior to drug administration, or recent participation in a clinical investigation that, in the opinion of the Investigator, would jeopardize subject safety or the integrity of the study results.
11. Received any type of live vaccine within 30 days prior to drug administration.
12. Use of medication within 30 days prior to drug administration.
13. On a special diet within 30 days prior to drug administration.
14. Have had a tattoo or body piercing within 30 days prior to drug administration.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
AUCt | From time 0 hours (prior to dosing), up to 48 or 72 hours post dose
  The area under the analyte concentration versus time curve, from time zero (0) to the time of the last measurable analyte concentration (t), as calculated by the linear up/log down variant of the trapezoidal method.
AUCinf | From time 0 hours (prior to dosing), up to 48 or 72 hours post dose
  The area under the analyte concentration versus time curve from time zero to infinity. AUCinf = AUCt + Ct/Kel, where Ct is the last measurable analyte concentration.
Cmax | From time 0 hours (prior to dosing), up to 48 or 72 hours post dose
  Maximum measured analyte concentration over the sampling period.
Tmax | From time 0 hours (prior to dosing), up to 48 or 72 hours post dose
  Time of the maximum measured analyte concentration over the sampling period.
Kel | From time 0 hours (prior to dosing), up to 48 or 72 hours post dose
  The apparent first-order elimination rate constant
Thalf | From time 0 hours (prior to dosing), up to 48 or 72 hours post dose
  The apparent elimination half-life

CONTACTS AND LOCATIONS:
Locations (1):
- Sandoz Investigational Site, Toronto, Ontario, Canada